CLINICAL TRIAL: NCT05709236
Title: Clinical Assessment of Maxillary Screw-retained Implant Prosthesis Fabricated From Digital Versus Conventional Full-arch Implant Impression: A Randomized Controlled Clinical Trial
Brief Title: Digital Versus Conventional Full-arch Implant Impression in Maxillary Screw- Retained Implant Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Wafaa Ibrahim, Associate Professor, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FODMRC/2022/00103
Record Dates: First submitted 2023-01-16; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Jaw, Edentulous
Keywords: edentulous; implant; Screw retained; Digital impression
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Completely edentulous maxillary arch digital impression (Experimental): treated with Maxillary screw-retained prosthesis with digital full-arch impression
  Interventions: Device: Maxillary screw-retained prosthesis
- Completely edentulous maxillary arch conventional impression (Active Comparator): treated with Maxillary screw-retained prosthesis with conventional full-arch impression
  Interventions: Device: Maxillary screw-retained prosthesis

INTERVENTIONS:
Device: Maxillary screw-retained prosthesis — Maxillary screw-retained prosthesis with conventional full-arch impression with conventional or digital impression

SUMMARY:
28 participants with edentulous maxillary arches were randomly selected and enrolled in two equal groups; Group I conventional impression group (CIG) and Group II Digital impression group (DIG). All patients were rehabilitated with maxillary screw-retained implant prosthesis retained by 6 implants. Prosthodontic complications and peri-implant MBL were registered at 6,12, and 24 months (m). Data was collected and statistically analyzed.

DETAILED DESCRIPTION:
Treatment sequence Pretreatment examination For all participants, diagnosis and treatment planning were performed. They were assessed clinically through oral examination by inspection and palpation, and radiographically using preoperative panoramic radiograph and cone beam computed tomography CBCT to evaluate bone morphology, bone height, bone density, and vertical as well as horizontal bone resorption.

New maxillary complete dentures were fabricated for all participants to serve as temporization and to perform prosthetically driven computer guided implant placement. Preoperative CBCT scan (i-CAT Visions; Imaging Sciences International, Hatfield, PA, USA) was performed for all participants using the newly fabricated dentures with extra oral ready-made radiopaque markers. The markers were placed in relation to the maxillary dentures laterals/canines position, first premolars position, and first molars position. The superimposition of these markers on the maxilla determines the potential implants sites. Implant planning was performed and a stereolithographic surgical guide was fabricated with 6 sleeves on these preplanned implants sites.

Surgical procedures Computer-guided surgery was performed; each participant of both groups received six axially placed implants (Neobiotech, South korea) in the preplanned implant positions in maxilla. The final insertion torque for implants was 40 N cm. Post-operative instructions were given for patients. Chlorhexidine mouth wash 0.2% was prescribed for two weeks.

Prosthetic procedures Patients of both groups were recalled after a healing period of soft and hard tissues of four months for second stage surgery. Transmucosal titanium abutments were screwed in after uncovering of the six implants. For the fabrication of the definitive prosthesis, two different approaches were implemented: conventional pick up versus digital impressions.

For group I patients (CIG), a conventional open tray full- arch implant impression was implemented to fabricate the definitive maxillary screw retained prosthesis. Six long impression transfers were screwed over the fixtures. Using a periapical radiographs the seating of the open-tray long impression copings was confirmed. Splinting of impression copings was performed using special resin (Duralay; Reliance Dental, Alsip, IL, USA) (Fig----). Conventional border molding of the custom open trays (Fig----) was performed, then light body vinyl polysiloxane (Imprint 3, 3M ESPE, St. Paul, MN, USA) was injected around the impression transfer (Fig---). The tray was then filled with a heavy body vinyl polysiloxane ((Imprint 3, 3M ESPE, St. Paul, MN, USA) and a conventional pick up impression was made. Implant analogues were then attached to the impression copings and stone models were pored to replicate the exact implant positions in the cast.

For group II patients (DIG), a digital full arch implant impression was utilized to fabricate the definitive maxillary screw retained prosthesis. A digital IOS (i-500®, Medit, Seoul, South Korea) and scan bodies (Neobiotech, South korea) replacing the traditional impression copings were used to capture accurately the implant fixtures. Splinting of the scan bodies was performed using the same technique employed for the impression transfers. The same experienced investigator performed the scanning of the splinted scan bodies applying the scanning stitching strategy 20.

Keeping the IOS light source parallel to the occlusal plane, scanning of the implants started from the distal left implant and then the IOS was moved toward the anterior right implant , and then moved back to the distal implant of the left quadrant, while tilting it palatally; followed by crossing the occlusal plan toward the buccal side.

The same scanning pathway was repeated from the starting scan point for each half. Inspection of the image and filling of the missing regions were performed by fast passages of the camera over the related areas.

Identical scanning of the other half was performed using consistent scanning procedures, from anterior left implant to the right distal implant of the contralateral quadrant. The software merges the two halves by applying a stitching algorithm which uses the shared area between the two anterior implants. Scanning of the soft tissues was then performed, and matching of the soft tissues and scan bodies of related components scans was achieved.

The "A.I. Scan Body Matching" feature was used in which the library data is aligned automatically with the scan data, minimizing the need to scan difficult-to-reach areas. Arranging and replacing that scan body data with the library data was completed to reproduce the position and angle of the implanted fixtures accurately.

Scanning of the opposing mandibular arch was accomplished using the same scanning procedures, followed by scanning of the buccal surface of the patients teeth in maximum intercuspation with the maxillary temporary denture.

The 3D scans created were then exported in STL format, uploaded and post processing accomplished. Accuracy of detail and correct occlusal relationship were evaluated for the virtual images and virtual models were created with dental implants in position.

Virtual digital creation of framework and prosthesis were performed using the CAD software (Exocad software, Darmstad, Germany) For both groups, milling of the definitive frameworks from titanium was performed in accordance with sending the rapid prototype model to the laboratory for the fabrication of the definitive prosthesis. The frameworks were seated and screwed to the implants fixtures and passive fit was ensured using Sheffield test. In none of the two groups the frameworks needed splitting and reassembling.

The prosthesis, set up for the esthetic trial placement, constituted by a framework and a suprastructure of esthetic material, has been refined in esthetics, function and in relation to soft tissues. After the esthetic and functional evaluation, the restoration is finalized, over the mesostructure the esthetic material has been added for the rebuilding of teeth with composite (NACERA HYBRID, DOCERAM Medical Ceramics GmbH, Dortmund, Germany) and soft tissues.

For both groups, the definitive prosthesis was cemented to the titanium mesostructured with a dual cure cement (Rely X Unicem, 3M, St. Paul, MN, USA), then positioning and screwing of the prosthesis onto the dental implants was accomplished and passive fit was ensured using the Sheffield test.

ELIGIBILITY:
Inclusion Criteria:

* patients with maxillary edentulous ridges opposing fully dentulous mandibular arch or with a minimum of six anterior teeth (canine to canine), and the utmost one or two premolar/molar missing in any quadrant
* patients with compromised facial/lip support seeking a fixed prosthesis for their edentulous maxilla
* having edentulous maxilla with adequate bone density and height to place six implants as assessed clinically and radiographically, and physically
* psychologically eligible patients for implants placement.

Exclusion Criteria:

* debarred medically compromised patients
* smokers
* patients suffering from parafunctional habits.

Ages: 56 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Number of events of prosthodontic complications | - 6 months, 12 months and 24 months
  For both groups, the prosthodontic complications of the maxillary screw-retained implant prosthesis were monitored and calculated during the twenty four months follow up period according to the following events: Loss of the cover of access hole, Framework fracture, Fractured acrylic resin, Prosthetic teeth fracture, Screw loosening of the abutment, Screw fracture of the abutment, Screw loosening of the prosthesis, Screw fracture of the prosthesis.

SECONDARY OUTCOMES:
Amount of marginal bone loss | 6 months, 12 months and 24 months
  Peri-implant MBL was assessed for the 6-implants in both groups at 6, 12, and 24 months using standardized digital peri-apical radiograph with long cone paralleling technique. Mesial and distal MBL relative to each implant shoulder was assessed in millimeters, and the mean was calculated and statistically estimated. Image analysis was performed using the Digora software (Digora phosphor plate reader; soredex, Tuusula, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa Ibrahim, PHD, Principal Investigator — Assoc. Prof.
Locations (1):
- Delta University for Science & Technology, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No